CLINICAL TRIAL: NCT03559244
Title: Investigating the Effects of Exercises in Addition to Dynamic Compression Brace in Patients With Pectus Carinatum: a Single Blinded Randomized Controlled Trial
Brief Title: Dynamic Compression Brace for Pectus Carinatum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 09.2018.328
Record Dates: First submitted 2018-05-20; First posted 2018-06-18 (Actual); Last update posted 2018-12-04 (Actual); Status verified 2018-07

CONDITIONS: Pectus Carinatum
Keywords: exercise; pectus carinatum; orthosis; dynamic compression brace
MeSH Terms: conditions — Pectus Carinatum; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Parallel group randomized controlled study
Who Masked: Outcomes Assessor
Masking Description: outcome assessor blinded to participants' allocated group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dynamic compression brace 8 hours (Experimental): Children with pectus carinatum who will wear dynamic compression brace 8 hours a day plus exercises for three weeks
  Interventions: Other: Dynamic compression brace; Other: Exercises
- Dynamic compression brace 23 hours (Experimental): Children with pectus carinatum who will wear dynamic compression brace 23 hours (except for bathing and sports activities) a day plus exercises for three weeks
  Interventions: Other: Dynamic compression brace; Other: Exercises
- Only exercises (Active Comparator): The children who are in wait in list for dynamic compression brace will receive only posture exercises, deep breathing exercises, exercises for manipulation and mobilization of ribs, and core exercises for three weeks
  Interventions: Other: Exercises

INTERVENTIONS:
Other: Dynamic compression brace — custom-fitted brace adjusts the pressure on the thoracic wall and enables lateral expansion of the thorax
  Arms: Dynamic compression brace 23 hours; Dynamic compression brace 8 hours
Other: Exercises — posture exercises, deep breathing exercises, exercises for manipulation and mobilization of ribs, and core exercises

SUMMARY:
Pectus carinatum (PC) is a deformity of the anterior chest wall which is a common pediatric condition, characterized by an idiopathic overgrowth of the costal cartilages resulting in protrusion of the sternum. Chest pain or discomfort, especially when lying in prone position, increased respiratory effort during exercise, scoliosis, impaired shoulders and kyphotic position are some of the physical signs and symptoms. Unlike pectus excavatum, PC is rarely associated with significant cardiopulmonary involvement except in severe cases. Pectus carinatum is not just a simple aesthetical problem. The effect of patient's self-esteem, body image and confidence can be variable and lead to significant deterioration in mental health. It can be responsible of physical signs and symptoms and also has significant psychological impact. Deformity and its psychological impact tend to worsen during pubertal rapid phases of growth and even during adult life. The management of pectus deformities used to include surgical techniques, however, recently compression brace which is a dynamic orthosis which is custom-fitted, rigid aluminum brace that is adjustable to any thoracic shape is widely applied instead of surgery. Pressure applied to the patient, in the most protruding area of the chest, needed to accomplish a proper shape of the thorax, the pressure of correction can be measured via a pressure measuring device in pounds per square inches (PSI). Treatment choices of surgery or bracing is determined according to pressure of correction and type of deformity. Surgical correction is indicated if the presence of chondro-manubrial type PC and pressure of correction > 10 PSI. Chest pain or discomfort, especially when lying in prone position, increased respiratory effort during exercise, scoliosis, impaired shoulders and kyphotic position are some of the physical signs and symptoms. Despite the fact that patients with PC have impaired posture, exercise intolerance and increased scoliosis occurrence, there is no consensus on the exercise program for patients with PC. Also, there is not enough scientific evidence about the wear time of orthosis. The aim of this study is to investigate the effects of exercises and compression brace in children with PC.

DETAILED DESCRIPTION:
Pectus carinatum (PC) is a deformity of the anterior chest wall which is a common pediatric condition, characterized by an idiopathic overgrowth of the costal cartilages resulting in protrusion of the sternum. There are two subtypes of PC: the chondro-gladiolar variant, which is the most common type, and presents with protrusion of the sternal body, and the chondro-manubrial variant, showing protrusion of the component of the sternum (manubrium). PC usually involves the lower sternal costal cartilages, pushing the sternum forwards and can be symmetrical (bilateral) or often asymmetrical (unilateral) with the right for some reason being more obviously affected. PC may occur as a solitary abnormality or in association with other genetic disorders or syndromes (eg, trisomy 18, Marfan syndrome, homocystinuria, Morquio syndrome, and Ehlers-Danlos syndrome). Of the musculoskeletal abnormalities, scoliosis is most frequently associated with PC.

Chest pain or discomfort, especially when lying in prone position, increased respiratory effort during exercise, scoliosis, impaired shoulders and kyphotic position are some of the physical signs and symptoms. Unlike pectus excavatum, PC is rarely associated with significant cardiopulmonary involvement except in severe cases. Pectus carinatum is not just a simple aesthetical problem. It can be responsible of physical signs and symptoms and also has significant psychological impact. Deformity and its psychological impact tend to worsen during pubertal rapid phases of growth and even during adult life. It has been demonstrated that patients with PC are at risk for a disturbed body image and reduced quality of life and many patients refer feelings of discomfort, shame, shyness, anxiety, and even depression.

The classical management of pectus deformities, both carinatum and excavatum, has been primarily surgical. Modification of the Ravitch technique involves resection of the deformed costal cartilages along with sternal osteotomy. Because the results of this technique resulted in worse cosmetic results, a new less invasive procedure, the Nuss procedure was developed. Nuss procedure includes remodeling of the chest wall cartilage with an internal support bar. These techniques have demonstrated the plasticity of the chest wall and led clinicians to hypothesize that carinatum defects would also remodel in response to chronic pressure, leading to a cosmetically superior, nonoperative technique: compression brace. Compression brace is a dynamic orthosis which is custom-fitted, rigid aluminum brace that is adjustable to any thoracic shape. Complications of brace use include uncommon (4.6%), mild and easy to resolve: back pain, hematoma and skin ulceration. Pressure of correction is the pressure applied to the patient, in the most protruding area of the chest, needed to accomplish a proper shape of the thorax. It is an indirect parameter of the chest wall's flexibility. It can be measured with a pressure measuring device in pounds per square inches (PSI). Some special designed braces contain a part in which pressure measuring device can be docked. This enables measuring of pressure of treatment. Pressure of treatment can be different from pressure of correction since skin breakdown occurs with corrections at high pressure.

In the Calgary protocol, wearing brace 23 hours a day during the correction phase until the development of the axial skeleton is completed and afterwards 8 hours of wear is recommended in the continuation phase.Martinez-Ferro et al developed pressure measuring device and special designed braces contain a part in which pressure measuring device can be docked. They suggested that patients with pressure of correction <10 should be braced. De Beer et al. also recommended the surgical treatment in the presence of chondro-manubrial type PC and pressure of correction > 10 PSI. However, recommendations are based on prospective or retrospective cohort studies other than randomized controlled trials which corresponds to low level of evidence.

Despite the fact that patients with PC have impaired posture, exercise intolerance and increased scoliosis occurrence, there is no consensus on the exercise program for patients with PC. Postural impairment aggravates psychological burden caused by disease itself. Patients with pectus carinatum may get benefit from exercises to improve posture. Also, disease itself or compression brace use may result in abdominal flare and increased lateral diameter of chest wall as an unwanted effect. Strengthening of abdominal muscles may prevent from abdominal flare. Strengthening of chest wall muscles, strengthening the pectoralis and sacrospinalis muscles as well as expanding the chest through deep breathing, strengthening core muscles including abdominal muscles, increasing flexibility of muscles, manipulation and mobilization of costae may lead improvements in the management of PC.

There is no consensus about exercises, and there is not enough scientific evidence about the wear time of orthosis. The existing treatment protocols are non-standardized protocols developed by the researchers of previous studies investigating the effectiveness of orthosis. Martinez-Ferro et al., the developer of the dynamic compression brace, recommends the daytime wear of orthosis for patients with low pressure of correction. They recommend duration of clothing to be shorter and the pressure of treatment should be kept lower in patients with high pressure of correction. However, every compression brace may not contain dock and pressure of treatment cannot be measured. In the present study we aimed to investigate the effects of exercises and compression brace in children with PC. Also, safety and feasibility of the orthosis will be evaluated. Patients with chondro-gladiolar, symmetrical or asymmetric, compressible PC (compression test positive) and with correction pressure ≤10 PSI, aged 5-18 years old will be included to study. They will be randomized to three groups using closed envelope system. All groups will be given exercises to strengthen the muscles of the respiratory muscles of the posture exercises, deep breathing exercises, ribs manipulation and mobilization exercises and core exercises for 1 hour a day, five days a week for 3 weeks. The first group will use the orthosis for 8 hours during the night and the second group for 23 hours except for sports activities, exercise and bath. The control group who will receive exercise therapy only will be selected from the wait-in list for the orthosis. Pectus carinatum protrusion, pressure of correction, anteroposterior and lateral diameter of thorax at the most protruded part of deformity, Haller index, Cobb and kyphosis angle, Pectus Evaluation Questionnaire will be assessed at before treatment and after treatment, 1 month and 3 months and 6 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male patients with pectus carinatum
2. Symmetric or asymmetric pectus carinatum
3. Compression test positive
4. Pressure of correction <10 PSI

Exclusion Criteria:

1. History of orthosis use
2. Chondro-manubrial pectus carinatum
3. Concomitant severe scoliosis (Cobb angle>20)
4. Having history of chronic disease
5. History of surgery for scoliosis or pectus carinatum

Ages: 5 Years to 20 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 27 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2018-12-02 (Actual); Study Completion 2018-12-02 (Actual)

PRIMARY OUTCOMES:
Pectus carinatum protrusion | Day 0
  distance from the point of maximum protrusion to the estimated normal level of chest wall
Pectus carinatum protrusion | 3 weeks
  distance from the point of maximum protrusion to the estimated normal level of chest wall

SECONDARY OUTCOMES:
T1 (external measurement of chest wall at the upper age of manubrium) | Day 0
  external measurement of the anterior chest wall using a thorax caliper at the upper edge of the manubrium
T1 (external measurement of chest wall at the upper age of manubrium) | 3 weeks
  external measurement of the anterior chest wall using a thorax caliper at the upper edge of the manubrium
T2 (external measurement of chest wall at Angulus Ludovici) | Day 0
  the external measurement of the anterior chest wall using a thorax caliper at the T2 point (Angulus Ludovici)
T2 (external measurement of chest wall at Angulus Ludovici) | 3 weeks
  the external measurement of the anterior chest wall using a thorax caliper at the T2 point (Angulus Ludovici)
T3 (external measurement of chest wall at the most protruded point from the chest wall) | Day 0
  the external measurement of the anterior chest wall using a thorax caliper at the T3 (the most protruded point from the chest wall)
T3 (external measurement of chest wall at the most protruded point from the chest wall) | 3 weeks
  the external measurement of the anterior chest wall using a thorax caliper at the T3 (the most protruded point from the chest wall)
Haller index | Day 0
  maximal transverse diameter/narrowest anteroposterior(AP) length of chest
Haller index | 3 weeks
  maximal transverse diameter/narrowest AP length of chest
Cobb angle | Day 0
  The angle between the lines which are drawn parallel to the upper endplate of the superior end vertebra and lower endplate of inferior end vertebra forms the Cobb angle (CA).
Cobb angle | 3 weeks
  The angle between the lines which are drawn parallel to the upper endplate of the superior end vertebra and lower endplate of inferior end vertebra forms the CA.
Kyphotic angle | Day 0
  the angle between the lines drawn along the upper endplate of T4 vertebra and lower endplate of T12 vertebra is calculated.
Kyphotic angle | 3 weeks
  the angle between the lines drawn along the upper endplate of T4 vertebra and lower endplate of T12 vertebra is calculated.
Pressure of correction | Day 0
  Pressure of correction (PC): an indirect parameter of the chest wall's flexibility. It is defined as the pressure applied to the patient, in the most protruding area of the chest, needed to accomplish a proper shape of the thorax.
Pressure of correction | 3 weeks
  Pressure of correction (PC): an indirect parameter of the chest wall's flexibility. It is defined as the pressure applied to the patient, in the most protruding area of the chest, needed to accomplish a proper shape of the thorax.
Pectus Evaluation Questionnaire patient form | Day 0
  The Nuss Questionnaire modified for Adults (NQmA) is a disease-specific health-related quality of life assessment tool for patients with pectus deformities.
Pectus Evaluation Questionnaire patient form | 3 weeks
  The Nuss Questionnaire modified for Adults (NQmA) is a disease-specific health-related quality of life assessment tool for patients with pectus deformities.
Pectus Evaluation Questionnaire parent form | Day 0
  The Nuss Questionnaire modified for Adults (NQmA) is a disease-specific health-related quality of life assessment tool for patients with pectus deformities.
Pectus Evaluation Questionnaire parent form | 3 weeks
  The Nuss Questionnaire modified for Adults (NQmA) is a disease-specific health-related quality of life assessment tool for patients with pectus deformities.
Thorax AP diameter measurement | Day 0
  Thorax AP diameter measurement with a thoracic caliper at the most protruded region
Thorax AP diameter measurement | 3 weeks
  Thorax AP diameter measurement with a thoracic caliper at the most protruded region
Thorax lateral diameter measurement | Day 0
  Thorax lateral measurement with a thoracic caliper at the most protruded region
Thorax lateral diameter measurement | 3 weeks
  Thorax lateral measurement with a thoracic caliper at the most protruded region

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Yuksel, Prof, Study Chair — Marmara University; Gulseren Akyuz, Prof, Study Director — Marmara University
Locations (1):
- Marmara University School of Medicine Department of Physical Medicine and Rehabilitation, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fokin AA, Steuerwald NM, Ahrens WA, Allen KE. Anatomical, histologic, and genetic characteristics of congenital chest wall deformities. Semin Thorac Cardiovasc Surg. 2009 Spring;21(1):44-57. doi: 10.1053/j.semtcvs.2009.03.001. PMID 19632563
- [Background] Martinez-Ferro M, Bellia Munzon G, Fraire C, Abdenur C, Chinni E, Strappa B, Ardigo L. Non-surgical treatment of pectus carinatum with the FMF(R) Dynamic Compressor System. J Vis Surg. 2016 Mar 17;2:57. doi: 10.21037/jovs.2016.02.20. eCollection 2016. PMID 29078485
- [Background] Kravarusic D, Dicken BJ, Dewar R, Harder J, Poncet P, Schneider M, Sigalet DL. The Calgary protocol for bracing of pectus carinatum: a preliminary report. J Pediatr Surg. 2006 May;41(5):923-6. doi: 10.1016/j.jpedsurg.2006.01.058. PMID 16677884
- [Background] de Beer SA, Gritter M, de Jong JR, van Heurn ELW. The Dynamic Compression Brace for Pectus Carinatum: Intermediate Results in 286 Patients. Ann Thorac Surg. 2017 Jun;103(6):1742-1749. doi: 10.1016/j.athoracsur.2016.12.019. Epub 2017 Mar 6. PMID 28274516
- [Background] Banever GT, Konefal SH, Gettens K, Moriarty KP. Nonoperative correction of pectus carinatum with orthotic bracing. J Laparoendosc Adv Surg Tech A. 2006 Apr;16(2):164-7. doi: 10.1089/lap.2006.16.164. PMID 16646710
- [Background] Lee RT, Moorman S, Schneider M, Sigalet DL. Bracing is an effective therapy for pectus carinatum: interim results. J Pediatr Surg. 2013 Jan;48(1):184-90. doi: 10.1016/j.jpedsurg.2012.10.037. PMID 23331813